CLINICAL TRIAL: NCT02259465
Title: A Randomised Controlled Trial of the Effect of the Low FODMAP Diet and Dietary Oligofructose on Gastrointestinal Form, Function and Microbiota in Healthy Volunteers
Brief Title: The Effect of the Low FODMAP Diet and Dietary Oligofructose on Gastrointestinal Form, Function and Microbiota
Acronym: FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SoM A14082014 FOG
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: microbiota; FODMAP; oligofructose; Magnetic Resonance Imaging; Metabolomics; Diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet; oligofructose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oligofructose (Active Comparator): Participants will be asked to follow the low FODMAP diet for a week, supplementing the diet with oligofructose, 7grams twice daily
  Interventions: Behavioral: low FODMAP diet; Dietary Supplement: Oligofructose
- Maltodextrin (Placebo Comparator): Participants will be asked to follow the low FODMAP diet for a week, supplementing the diet with maltodextrin, 7grams twice daily
  Interventions: Behavioral: low FODMAP diet; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Behavioral: low FODMAP diet — Participants will attend a one-hour group session on how to follow the low FODMAP diet, run by a dietitian trained in the diet. They will be asked to follow the diet for 7 days while keeping a food diary.
Dietary Supplement: Oligofructose — Participants will supplement their diet with 7 grams of OF twice daily for the week that they follow the low FODMAP diet.
  Other Names: OraftiP95, OF
  Arms: Oligofructose
Dietary Supplement: Maltodextrin — Participants will supplement their diet with 7 grams of maltodextrin twice daily for the week that they follow the low FODMAP diet.
  Arms: Maltodextrin

SUMMARY:
Some carbohydrates, complex sugars, which are found in grains, fruit and vegetables, cannot be digested by humans. When eaten they pass through the small bowel to the large bowel, or colon. Some bacteria that live in the colon are able to digest these carbohydrates, and use them as an energy source. This releases energy that humans can absorb, and may have other effects on health as well. The process also releases gases such as hydrogen and methane into the colon, which will eventually be released as flatulence.

There is some evidence in animals, and humans, that changing the carbohydrate content of the diet may increase the numbers of bacteria in the colon that can use this energy source. Recent work has looked at how changes in colon bacteria and carbohydrate in the diet affect transit, the speed at which food and stool moves through the stomach and bowels.

This undergraduate project will use techniques in Magnetic Resonance Imaging developed in Nottingham to investigate how a prolonged change in dietary carbohydrate might affect speed of transit through the bowel and gas production in the colon, and whether there is any immune reaction to the carbohydrate from the bowel wall.

DETAILED DESCRIPTION:
Oligofructose (OF) is a fructose- based oligosaccharide and defined in the European Union as a dietary fibre. Enzymatically derived from the longer chain inulin in chicory, it is commonly used in processed food to improve mouth feel in fat-free products. OF is poorly digested and absorbed in the small bowel so passes to the colon where it is fermented by the bacteria usually resident in the colon, termed the microbiota. This process produces gases such as hydrogen and sometimes methane, and short-chain fatty acids (SCFAs) which have a variety of roles including nutrition to colonocytes, immunological effects and modulation of intestinal motility. Its presence in the colon alters the composition of the microbiota, with reported potential benefits to health, leading to its description as a 'prebiotic'.

Recently, however, such poorly digested carbohydrates grouped together by the term FODMAP (fermentable oligo-, di-, mono-saccharides and polyols) have been proposed to exacerbate symptoms of irritable bowel syndrome (IBS) such as abdominal discomfort and bloating. Dietary exclusion of foods containing FODMAPs, such as wheat, dairy and certain fruit and vegetables, has been proposed as a treatment for IBS, with some evidence to support this. FODMAPs are thought to induce symptoms either by drawing water into the small bowel by osmosis, or through gaseous distension of the large bowel or a combination of these along with metabolite effects on motility.

The Nottingham GI MRI group has been at the forefront of elucidating the actual effects of FODMAPs on gastrointestinal (GI) physiology. We have published techniques to measure small bowel water content, colonic volume and gas volume and whole gut transit time. We have recently demonstrated that a single, large (40g) dose of inulin leads to an increase in colonic volume, mainly through an increase in colonic gas. Such a dose is beyond the usual range of dietary variation, however. Last year we piloted a model more similar to dietary practice. Participants supplemented their usual diet with 5g OF twice daily for a week. The most striking result was an 18% increase in fasting colonic volume. This could not be explained by changes in colonic gas and may represent proliferation, and increased mass, of the microbiota. That study was an open label, uncontrolled case series so we now wish to test the hypothesis in a double-blind, randomised controlled trial. For explanatory purposes we will also measure whole gut transit, colonic gas volume and hydrogen and methane expired in the breath. For exploratory purposes we will also collect stool and urine samples to allow assessment of the effect on microbiota and their metabolic output.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Able to give informed consent

Exclusion Criteria:

* Self-declared vegetarian, vegan or kosher/ halal diet who cannot eat carmine red dye
* Pregnancy declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function
* A positive diagnosis of irritable bowel syndrome based on the Rome III criteria questionnaire
* Reported history of previous resection of the oesophagus, stomach or intestine (excluding appendix)
* Intestinal stoma
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Will not limit alcohol intake to ≤ 35 units/ week and ≤ 8 units per day during trial
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Antibiotic or prescribed probiotic treatment in the past 8 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in colonic volume | one week
  Percentage change from baseline in fasting colonic volume after one week of intervention, as measured by Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Change in whole gut transit time | one week
  Change in whole gut transit time (WGTT) after one week of intervention, as determined by Weighted Average Position Score (WAPS) of MRI transit markers 24 hours after ingestion
Change in colonic gas volume | one week
  Percentage change in fasting colonic gas volume after one week of intervention, as measured by MRI
Change in fasting breath hydrogen | one week
  Change in fasting breath hydrogen concentration after one week of intervention, measured in parts per million
Change in fasting breath methane | one week
  Change in fasting breath methane concentration after one week of intervention, measured in parts per million

OTHER OUTCOMES:
Change in urinary metabolites | one week
  Exploratory work to assess change in urinary metabolite concentrations after one week of intervention
Change in faecal microbiota | one week
  Exploratory work to assess change in faecal microbiota concentrations after one week of intervention
Change in faecal short-chain fatty acids | one week
  Exploratory work to assess change in faecal short-chain fatty acid concentrations after one week of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD FRCP, Study Chair — University of Nottingham; Giles AD Major, BMBCh MRCP, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre, Nottingham, United Kingdom

REFERENCES:
- See also: Related Info — http://www.nddcbru.org.uk
- See also: Related Info — https://www.facebook.com/UoN.Gastrointestinal.MRI